CLINICAL TRIAL: NCT05683288
Title: Comparison of the Efficiency of Instrument Assisted Soft Tissue Mobilization and Myofascial Release Techniques in Individuals With Chronic Neck Pain
Brief Title: Short and Long Time Effects of IASTM and Myofascial Release Techniques in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUH7
Record Dates: First submitted 2022-12-28; First posted 2023-01-13 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2022-12

CONDITIONS: Chronic Neck Pain
Keywords: Chronic Neck Pain; Disability; Pain
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IASTM (Experimental): EYYDM will be applied to the upper trapezius and sternocleideomastoid muscles of the participants for 90 seconds, with a frequency of 60 beats per minute. The instruments will be applied to the soft tissue at 30º-60º angles with multidirectional strokes ("stroking") movements.
  Interventions: Other: IASTM
- Myofascial Release (Experimental): Basic movements will be used in the rectus capitis, sternocleidomastoideus, hyoid region and upper trapezius regions within the scope of myofascial release application. The application will take 3 minutes for each region.
  Interventions: Other: Myofascial Release
- Control (Experimental): It will include 250W infrared application on the cervical region from 50cm away for 15 minutes and TENS application for 20 minutes at 80Hz frequency with 150ms current transit time, home exercise program.
  Interventions: Other: 250W infrared application; Device: TENS; Other: Home exercise

INTERVENTIONS:
Other: IASTM — IASTM will be applied to the upper trapezius and sternocleidomastoid muscles of the participants for 90 seconds, with a frequency of 60 beats per minute.
  Arms: IASTM
Other: Myofascial Release — Basic movements will be performed for 3 minutes in the rectus capitis, sternocleidomastoideus, hyoid region and upper trapezius regions.
  Arms: Myofascial Release
Other: 250W infrared application — For 15 minutes, 250W infrared application will be applied on the cervical region from a distance of 50 cm
  Arms: Control
Device: TENS — TENS will be applied for 20 minutes at 80Hz frequency, with a current transit time of 150ms.
  Arms: Control
Other: Home exercise — Cervical strengthening and stretching exercises five days a week will given
  Arms: Control

SUMMARY:
The aim of this study is to determine whether EYYDM and myofascial applications have short and long-term effects on pain and disability in individuals diagnosed with chronic neck pain.

DETAILED DESCRIPTION:
Participants will be randomly assigned to IASTM, myofascial release and control groups. In addition to conventional treatment, IASTM and myofascial release groups will be treated twice a week for 4 weeks. Conventional treatment will be applied to the control group for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of chronic neck pain,
* To have given at least 3 values to the pain with the Numerical Pain Scale
* having bilateral muscle spasms in the cervical region

Exclusion Criteria:

* those who are taking any analgesic medication,
* those with acute injury or infection,
* those with open wounds,
* osteoporosis,
* fracture,
* hematoma,
* those with acute cardiac, liver and kidney problems,
* those with connective tissue disease,
* rheumatoid arthritis, osteoarthritis,
* cancer,
* those with circulation problems,
* those with peripheral vascular disease,
* epilepsy,
* history of surgery in the cervical region

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cervical Pain assessed by Numeric Pain Scale. | Baseline, 4 weeks
  Pain will be evaluated with a 10-point Likert Numerical Pain Scale. 0 means no pain, 10 means unbearable pain.

SECONDARY OUTCOMES:
Change from Baseline Cervical Disability assessed by Neck Disability Index | Baseline, 4 weeks
  Cervical Disability will be evaluated with Neck Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)